CLINICAL TRIAL: NCT02436733
Title: EORTC Randomized Phase II Study of Pleurectomy/ Decortication (P/D) Preceded or Followed by Chemotherapy in Patients With Early Stage Malignant Pleural Mesothelioma
Brief Title: Pleurectomy/ Decortication (P/D) Preceded or Followed by Chemotherapy in Patients With Early Stage MPM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1205
Record Dates: First submitted 2015-04-21; First posted 2015-05-07 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: pleural mesothelioma; phase II; randomized; surgery; chemotherapy; feasibility
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cerebral Decortication; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate pleurectomy/decortication (Experimental): immediate P/D followed by three cycles of pemetrexed 500mg/m2 IV and cisplatin 75 mg/m2 IV, both drugs given on day 1, every three weeks for non-progressing patients
  Interventions: Procedure: pleurectomy/decortication; Drug: Pemetrexed/Cisplatin
- Delayed pleurectomy/decortication (Active Comparator): three cycles of pemetrexed 500mg/m2 IV and cisplatin 75 mg/m2 IV, both drugs given on day 1, every three weeks followed by P/D, for non-progressing patients.
  Interventions: Procedure: pleurectomy/decortication; Drug: Pemetrexed/Cisplatin

INTERVENTIONS:
Procedure: pleurectomy/decortication — Lung sparing procedures consist of the resection of the pleura without removing the lung
  Other Names: P/D
Drug: Pemetrexed/Cisplatin — On day 1 of each cycle, pemetrexed 500 mg/m2 should be administered as IV infusion followed by cisplatin 75 mg/m2 as IV.
  Other Names: CisPem

SUMMARY:
This is a multicenter, randomized, 1:1, non-comparative phase II trial. Patients with early stage MPM will be randomized between Arm A: immediate P/D followed by three cycles of chemotherapy (pemetrexed 500mg/m2 and cisplatin 75 mg/m2, both drugs given on day 1, every three weeks) Arm B: three cycles of chemotherapy (same regimen) followed by P/D, for non-progressing patients

DETAILED DESCRIPTION:
This is an academic led, multicenter, randomized, 1:1, non-comparative phase II trial. Patients with early stage MPM will be randomized between

* Arm A - immediate surgery: immediate P/D followed by three cycles of chemotherapy (pemetrexed 500mg/m2 and cisplatin 75 mg/m2, both drugs given on day 1, every three weeks) for non-progressing patients
* Arm B - delayed surgery: three cycles of chemotherapy (same regimen) followed by P/D, for non-progressing patients.

A maximum of four weeks (±2 weeks) will be allowed between the baseline tumor assessment and the start of treatment (surgery or chemotherapy). Randomization should be done as soon as possible after baseline tumor assessment.

The primary objective of the study is to investigate the feasibility of immediate P/D followed by cisplatin/pemetrexed chemotherapy or deferred P/D after cisplatin/pemetrexed chemotherapy in patients with early stage MPM.

The results of this study will allow the LCG to take one of the arms further to a comparative study with either no surgery or EPP as control arm. The choice of the comparator will depend on the result of a parallel ongoing randomized study in the UK, comparing P/D with no surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, with pathologically proven malignant pleural mesothelioma. All histological subtypes are accepted.
* Stage cT1-3, N0-2, M0 according to UICC TNM classification. FDG-PET-CT scan showing absence of M1, N3, supraclavicular and coeliac node involvement is required. No clinical invasion of mediastinal structures (heart, aorta, spine, esophagus, etc.) and no widespread chest wall invasion (T4) are acceptable. Focal chest wall lesions are acceptable.
* No prior treatment of any kind for mesothelioma is allowed, especially prophylactic track irradiation after diagnostic procedures.
* WHO performance status 0-1
* Fit to receive chemotherapy and undergo a pleurectomy/ decortication with optional removal of hemidiaphragm and pericardium.
* No history of other malignancy within the last three years, except for carcinoma in situ of the cervix or basal cell or spinocellular carcinoma of the skin.
* No pre-existing peripheral sensory or motor neuropathy > grade I according to CTCAE v4.0
* No clinically significant pleural effusion that cannot be managed with thoracentesis or pleurodesis (according to institutional practice). If pleurodesis is considered, it should be done before randomization.
* Adequate organ function Women of child bearing potential must have a negative serum (or urine) pregnancy test within 3 days prior to the start of chemotherapy/surgery. Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least three months after the last study treatment.

Before patient registration written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria

• Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease; wound healing disorders; ulcers; or bone fractures, known infection with HIV, active hepatitis B and/or hepatitis C virus).

significant cardiovascular morbidity (assessed by cardiologist) precluding surgery

* Major surgical procedure or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery (other than P/D) during the course of study treatment.
* History of receiving any investigational treatment within 28 days of randomization.
* History of intolerance to pemetrexed and/or cisplatin.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-09-20 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Rate of success to complete the full treatment | 20weeks
  A patient is considered to be a "treatment success" if he/she meets all of the following criteria:
  1. Patient has received the full protocol treatment, defined as 3 cycles of pemetrexed and cisplatin (allowing for the dose adjustments described in section 5.3), preceded/followed by pleurectomy/decortication (P/D) (as described in section 5.3).
  2. Patient alive and has no evidence of progression/relapse at week 20 (±2 weeks) after the first day of starting protocol treatment (either chemotherapy or P/D).
  3. Patient has no persisting grade 3-4 treatment side-effects (CTCAE V 4.0) at week 20 (±2 weeks) after the first day of starting protocol treatment (either chemotherapy or P/D)

SECONDARY OUTCOMES:
Loco-regional failure free survival | 6 months
  Loco-Regional Failure Free Survival (LRFFS) is defined as the time interval between the date of randomization and the date of relapse in hemithorax or mediastinum or death, whichever comes first
Overall survival | 15 months
  the time interval between the date of randomization and the date of death of any cause
Treatment side-effects | 36 weeks
  Treatment side-effects will be assessed for all patients and graded per CTCAE category upon occurrence of the event. The investigator will assess whether those events are surgery or/and drug related (no reasonable possibility, reasonable possibility) and this assessment will be recorded in the database for all adverse events. Surgical side effects during the perioperative period will be scored according to the Clavien-Dindo Classification of Surgical Complications as an exploratory approach.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Meerbeeck, Pr., Principal Investigator — UZ Antwerpen, Belgium
Locations (4):
- Belgium (2):
  - UZ Antwerpen, Antwerp
  - UZ Gent, Ghent
- Netherlands (2):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Erasmus MC Hospital, Rotterdam

IPD SHARING:
Plan to Share IPD: No